CLINICAL TRIAL: NCT05050227
Title: Improving Depression Management in Primary Care (CDA 19-108)
Brief Title: Improving Depression Management
Acronym: IDMPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDX 21-004; IK2HX002867 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: depression; primary health care; cognitive behavioral therapy; veterans
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cCBT Enhanced Collaborative Care (Experimental): Participants in the intervention arm will receive computerized cognitive behavioral therapy (cCBT) supported by a depression care manager in addition to the usual care provided.
  Interventions: Behavioral: cCBT Enhanced Collaborative Care
- Usual Care (Active Comparator): Participants in the usual care arm will receive the usual care provided as described below.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: cCBT Enhanced Collaborative Care — Computerized CBT (cCBT) will be delivered supported by a depression care manger who will facilitate access to cCBT, promote and monitor cCBT use, reinforce CBT concepts (during outside CBT session "homework"), and monitor mental health symptoms for each participant.
  Arms: cCBT Enhanced Collaborative Care
Behavioral: Usual Care — Primary Care Provider supported usual care typically includes medication prescription and referrals to specialty mental health, including Primary Care - Mental Health Integration services.
  Arms: Usual Care

SUMMARY:
Depression is disabling and affects one in five Veterans. VA's Primary Care-Mental health Integration (PC-MHI) enables specialists to support medication treatment in primary care, but timely and sufficient access to psychotherapy is unattainable despite Veteran preference for psychotherapy. This study aims to close the gap in psychotherapy access for VA primary care patients with depression by adapting and pilot testing PC-MHI collaborative care models to improve uptake of computerized cognitive behavioral therapy (cCBT).

DETAILED DESCRIPTION:
Background: VA's Primary Care-Mental Health Integration (PC-MHI) is rooted in evidence-based collaborative care models, where care managers, mental health specialists, and primary care providers jointly treat depression in primary care. While PC-MHI enabled specialists to support medication treatment in primary care, timely and sufficient access to psychotherapy is unattainable. Alternative therapy modalities are needed.

Significance/Impact: Depression is disabling and affects one in five Veterans. Psychotherapy is preferred by Veterans, but fraught with multilevel barriers (e.g., staff availability, patient travel to clinic, limited clinic hours). Without enhancing existing PC-MHI models to enable better primary care patient access to effective psychotherapies, Veteran engagement in depression treatment is unlikely to improve.

Innovation: This study aims to close the gap in psychotherapy access for VA primary care patients with depression by adapting PC-MHI collaborative care models to improve uptake of computerized cognitive behavioral therapy (cCBT). cCBT is accessible 24/7 via the internet and has effectively treated depression in more than 30 trials. With modest specialist support, it is non-inferior to face-to-face psychotherapy. PC-MHI can facilitate Veteran uptake of cCBT, using an evidence-based collaborative care model to provide the follow-up care management and mental health specialist back-up that characterizes the most effective cCBT trials.

Specific Aims/Methodology: To pilot test the feasibility, acceptability, and potential effects of cCBT-enhanced collaborative care on Veterans' depression symptoms and related outcomes in VA Greater Los Angeles Healthcare System. A pilot randomized controlled trial (RCT) will be conducted to examine feasibility, acceptability, and potential effects on depression, patient activation, and health-related quality of life in VA primary care patients with depression receiving either (1) cCBT-enhanced collaborative care (n=37) or (2) usual care (n=37) in West Los Angeles VA, from baseline to 3-months (post-intervention).

Next Steps/Implementation: Adapting PC-MHI's collaborative care model to incorporate cCBT can improve access to psychotherapy and engage the ~400,000 untreated Veterans with depression who prefer psychotherapy, especially OIF/OEF/OND Veterans seeking care that is convenient.

ELIGIBILITY:
Inclusion Criteria:

* Have access to computer (mobile or desktop), internet, telephone, and email
* Able to read English text on a computer screen
* Score 10 or higher on the PHQ-9

Exclusion Criteria:

* Have moderate-high suicide risk (e.g., suicide flag) or active suicidality
* Have other serious mental illness (e.g. bipolar disorder, psychosis)
* Have medical disorder that would prevent/interfere with participation (e.g. dementia/cognitive impairment, terminal illness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 37 self-identified male individuals and 37 self-identified female individual will be enrolled in the study
Enrollment: 57 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda B Leung, MD MPH PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Started | 29 | 28
Completed | 21 | 21
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (17.6) | 49.8 (15.1) | 49.9 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 21 | 19 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 9 | 17
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 8 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 28 | 57
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The minimum score is 0, the maximum is 27. A higher score indicates a worse outcome (i.e. more severe depression symptoms).
  units on a scale | 15.4 (4.9) | 14.6 (5.2) | 15.1 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) is a scale commonly used to measure and categorize depression symptoms. It is already administered as part of routine primary care at our study site. The minimum score is 0, the maximum is 27. A higher score indicates a worse outcome (i.e. more severe depression symptoms).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | 12.6 (5.2) | 15.2 (5.1)

2. Secondary Outcome: PROMIS Global Health
Description: The 10-item PROMIS Global Health assesses health-related quality of life and is summarized into "physical health" (physical functioning, pain, fatigue) and "mental health" (emotional problems, social functioning). Raw scores are summed (minimum score for either physical health or mental health=4, maximum score for either =20) and converted to a t-score by using a conversion table (minimum t-score for physical health=16.2, maximum =67.7; minimum t-score for mental health=21.2, maximum =67.6). A score of 50, with a standard deviation of 10, is the average for the United States general population. For both the physical and mental health, a higher score indicates a better outcome (i.e., better health). For physical health, a score of 35 or less is reflective of "poor" physical health, and 36-42 of "fair". Similarly, for mental health, a score of 29 or less is reflective of "poor" mental health, 29-40 of "fair".
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Number analyzed (Participants) | 21 | 21
t-score
  Physical Health | 38.3 (7.1) | 38.7 (8.4)
  Mental Health | 36.9 (6.1) | 38.2 (6.5)

3. Secondary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: The 7-item Generalized Anxiety Disorder (GAD-7) is among the most commonly used and best validated anxiety measures in primary care settings. The minimum score is 0, the maximum is 21. Higher scores indicate a worse outcome (i.e., more severe anxiety). For reference: scores of 0-4=minimal anxiety, 5-9=mild anxiety, 10-14=moderate anxiety, and 15-21=severe anxiety.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | 9.6 (5.8) | 10.6 (5.2)

4. Secondary Outcome: Patient Activation Measure (PAM)
Description: The 13-item Patient Activation Measure (PAM) will be used to assess an individual's knowledge, skill, and confidence for self-management. The minimum score is 0, the maximum is 100. Higher scores indicate a better outcome (i.e., higher patient activation).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | 37.5 (4.2) | 38.6 (5.4)

5. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-reported measure that will be used to assesses PTSD symptoms and symptom change. The minimum score is 0, the maximum is 80. Higher score indicate a worse outcome (i.e., more severe PTSD symptoms).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | 30.1 (19.5) | 34.0 (16.7)

6. Secondary Outcome: Behavioral Activation for Depression Scale (BADS-SF)
Description: The 9-item Behavioral Activation for Depression Scale (BADS-SF) will also be used to examine behavioral activation as an intermediary to depression symptomatology outcomes. The minimum score is 0, the maximum is 54. Higher scores indicate a better outcome (i.e., higher activation).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | 21.4 (9.1) | 22.6 (7.8)

7. Other Pre Specified Outcome: Treatment Engagement
Description: Treatment engagement will be conceptualized as the number of cCBT sessions completed. The minimum number of sessions is 0 and the maximum is 11. A higher number indicates more cCBT sessions completed, but isn't indicative of a better or worse outcome.
Time Frame: 3-months
Population: Usual care participants were not given the opportunity to use the cCBT program.
Measure: Mean (Standard Deviation); unit: number of sessions
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
Number analyzed (Participants) | 29 | 0
number of sessions | 6.7 (4.9) |

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | cCBT Enhanced Collaborative Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT05050227/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT05050227/ICF_000.pdf